CLINICAL TRIAL: NCT06855719
Title: Effectiveness of a Multimodal Intervention With Simulation for Learning Home Health Nursing Care of Patients With Multimorbidity and Heart Failure: A Randomized Controlled Trial
Brief Title: Effectiveness of a Multimodal Intervention With Simulation for Learning Home Health Nursing Care of Patients With Multimorbidity and Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, Antonio Jesús Marín Paz, Principal Investigator, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 087_2024
Record Dates: First submitted 2025-02-22; First posted 2025-03-04 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Multimorbidity; Heart Failure
Keywords: High Fidelity Simulation Training; Patient Simulation; Home Health Nursing; Primary Care Nursing; Family Nursing; Nursing Education Research; Students, Nursing; Education, Nursing
MeSH Terms: conditions — Heart Failure | interventions — Multimorbidity

STUDY DESIGN:
Intervention Model Description: This study is a parallel group-randomized controlled trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: To guarantee the objectivity and impartiality of the study, masking will be performed, which implies that the random assignment of the participants to the groups, the evaluation of the performance of the nursing students in the simulations in the pretest and posttest, and the subsequent statistical analysis of the data will be performed by researchers external to the study. Also, the evaluators of the simulations and the data analyst will not know the assignment of the participants to the Control and Experimental groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Students will receive simulation training, which will be evaluated through individual and group debriefing sessions. They will also have access to their recording simulations for autonomous learning. They will learn the protocols and current scientific evidence on the care of multipathologic patients with heart failure.
  Interventions: Other: Training in high-fidelity simulation and knowledge of care protocols in patients with multimorbidity and heart failure
- Control Group (No Intervention): Students will receive only theoretical teaching about primary health care in nursing.

INTERVENTIONS:
Other: Training in high-fidelity simulation and knowledge of care protocols in patients with multimorbidity and heart failure — Participants will perform an individual simulation as nurses related to the patient profile in their home (pretest and postest). After each simulation, each participant will receive a recording of their simulation, and both individual and group debriefings will be conducted. In addition, they will be trained in scientific evidence and international and national protocols regarding the care of these patients in the context of home health nursing.
  Arms: Experimental Group

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of a multimodal intervention with high-fidelity simulations on home health nursing in improving the care of multipathological patients with heart failure in nursing students. The main questions it aims to answer are:

* Does using validated simulation scenarios on multipathological patients with heart failure improve care competencies in nursing students?
* Does knowledge of scientific evidence and healthcare protocols improve nursing students' performance in the simulator?

Researchers will compare a multimodal intervention with high-fidelity simulations on home health nursing to conventional intervention (theoretical teaching) to see if nursing students better learn competencies related to the care of patients with multimorbidity and heart failure during the home health nursing.

Participants will:

* Experience simulations on validated simulation scenarios on multipathological patients with heart failure (All participants).
* Reflect on the intervention performed on the simulator through individual and group debriefings (Experimental Group).
* Learn about the main scientific evidence and international and national protocols related to comorbidities and health failure (Experimental Group).

ELIGIBILITY:
Inclusion Criteria:

* Nursing students enrolled in the subject "Family and Community Nursing I".

Exclusion Criteria:

* Lack of attendance since the beginning of the course.
* Failure to follow the instructions of the instructors during the course of the study.
* Voluntary withdrawal from the study during the study or declaring non-participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Learning | From enrollment to the end of intervention at 4 weeks.
  Learning will be analyzed through nursing students' performance during the simulations. Two independent observers with experience in tesching simulation will evaluate each simulation (pretest and posttest) through a validated checklist for each simulation scenario. The checklist evaluates the following aspects: (1) assessment of people and observation of the home (4 items), (2) nursing intervention (5 items), and (3) transversal competencies related to greeting, farewell, and communication skills (5 items). Each item will be evaluated by a dichotomous response (Yes/No) and a final overall evaluation (0-10 points). The observers' degree of agreement will be determined by Cohen's kappa.
Empathy | From enrollment to the end of treatment at 4 weeks.
  Empathy toward patients presenting with pluripathologies and heart failure is essential for providing professional care. The general measure of the students' empathy level was measured by the Spanish version of the Jefferson Scale of Empathy, student version (JSE-S), with a Cronbach's alpha coefficient of 0.90. The JSE-S is a 20-item instrument specifically developed to measure empathy in health profession education and patient care for administration to health profession students and practitioners. Items are answered on a 7-point Likert-type scale (1 = Strongly Disagree, 7 = Strongly Agree). Half of the items are positively worded and directly scored, and the other half are negatively worded (reverse scored). The total score are range from 20 to 140, where a higher score indicates greater empathy.

SECONDARY OUTCOMES:
Self-confidence in learning | From enrollment to the end of treatment at 5 weeks
  Immediately after the simulation was performed. This will be measured using the Student Satisfaction and Self-Confidence in Learning (SCLS) scale. The scale is based on a five-point Likert scale, ranging from "strongly disagree" to "strongly agree." The scores that can be obtained range from 13 to 65 points and were validated with a Cronbach's alpha of 0.90.
Quality of simulations | From enrollment to the end of treatment at 5 weeks
  After the individual and group debriefings. The Educational Practices Questionnaire (student version) (EPQ) will be used. It consists of 16 items, assessed on two 5-point scales. Each item assessed quality and importance. The questionnaire is validated with Cronbach's alphas of 0.86 and 0.91 for the scales respectively.
Satisfaction on simulations | From enrollment to the end of treatment at 5 weeks
  After the individual and group debriefings. For this purpose, the High Fidelity Clinical Simulation satisfaction scale in students (ESSAF) will be used. This scale contains 33 statements answered on a 5-point Likert-type scale, with a minimum score of 1 (strongly disagree) to 5 (strongly agree). The 33 items are grouped into 8 factors or dimensions of student perception of the simulation clinic: "Usefulness", "Characteristics of cases and applications", "Communication", "Perceived performance", "Increased self-confidence", "Relationship between theory and practice", "Facilities and equipment" and "Positive aspects". It is validated with a Cronbach's alpha of 0.857.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Algeciras, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data related to the research, including those related to the participants (preserving anonymity), will be registered in a public data repository (institutional or international).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: * Study Protocol: February 2025 - March 2025.
  * SAP: March 2025 - December 2025.
  * ICF: March 2025 - December 2025.
  * Analytic Code: March 2025 - December 2025.
Access Criteria: Researchers and anyone will be able to access the data through a public repository and supplementary material if the study is published in an academic journal.

REFERENCES:
- [Background] Zeidi IM, Morshedi H, Alizadeh Otaghvar H. A theory of planned behavior-enhanced intervention to promote health literacy and self-care behaviors of type 2 diabetic patients. J Prev Med Hyg. 2021 Jan 14;61(4):E601-E613. doi: 10.15167/2421-4248/jpmh2020.61.4.1504. eCollection 2020 Dec. PMID 33628967
- [Background] Turen S, Enc N. A comparison of Gordon's functional health patterns model and standard nursing care in symptomatic heart failure patients: A randomized controlled trial. Appl Nurs Res. 2020 Jun;53:151247. doi: 10.1016/j.apnr.2020.151247. Epub 2020 Mar 5. PMID 32451005
- [Background] Villalba NL, Ballesteros BC, Alvarez LP, Mainar PD, Sanchez AN, Martinez JM, Manuel EC, Bailon MM. [Predictive factors of early readmission and mortality in patients with heart failure hospitalized in the Department of Internal Medicine of the San Carlos University Hospital, Spain]. Pan Afr Med J. 2019 Dec 17;34:202. doi: 10.11604/pamj.2019.34.202.17356. eCollection 2019. French. PMID 32180876
- [Background] Skou ST, Mair FS, Fortin M, Guthrie B, Nunes BP, Miranda JJ, Boyd CM, Pati S, Mtenga S, Smith SM. Multimorbidity. Nat Rev Dis Primers. 2022 Jul 14;8(1):48. doi: 10.1038/s41572-022-00376-4. PMID 35835758
- [Background] Santos GC, Liljeroos M, Dwyer AA, Jaques C, Girard J, Stromberg A, Hullin R, Schafer-Keller P. Symptom perception in heart failure - Interventions and outcomes: A scoping review. Int J Nurs Stud. 2021 Apr;116:103524. doi: 10.1016/j.ijnurstu.2020.103524. Epub 2020 Jan 10. PMID 32063295
- [Background] Jara Jara V, Sambuceti Nunez C. Clinical Simulation in Nursing: A Scale to Evaluate Satisfaction and Self-Confidence in Learning. Stud Health Technol Inform. 2018;250:89-90. PMID 29857393
- [Background] Merrou S, Baslam A, Idrissi Jouicha A, Ouhaz Z, El Adib AR. Blended learning and simulation in nursing education: A quasi-experimental study on a nursing institute. J Educ Health Promot. 2023 Sep 29;12:303. doi: 10.4103/jehp.jehp_72_23. eCollection 2023. PMID 38023106
- [Background] Martinez-Arce A, Rodriguez-Almagro J, Velez-Velez E, Rodriguez-Gomez P, Tovar-Reinoso A, Hernandez-Martinez A. Validation of a short version of the high-fidelity simulation satisfaction scale in nursing students. BMC Nurs. 2023 Sep 28;22(1):344. doi: 10.1186/s12912-023-01515-2. PMID 37770843
- [Background] Fernandez-Gutierrez M, Bas-Sarmiento P, Del Pino-Chinchilla H, Poza-Mendez M, Marin-Paz AJ. Effectiveness of a multimodal intervention and the simulation flow to improve empathy and attitudes towards older adults in nursing students: A crossover randomised controlled trial. Nurse Educ Pract. 2022 Oct;64:103430. doi: 10.1016/j.nepr.2022.103430. Epub 2022 Aug 22. PMID 36122493
- [Background] Fegran L, Ten Ham-Baloyi W, Fossum M, Hovland OJ, Naidoo JR, van Rooyen DRM, Sejersted E, Robstad N. Simulation debriefing as part of simulation for clinical teaching and learning in nursing education: A scoping review. Nurs Open. 2023 Mar;10(3):1217-1233. doi: 10.1002/nop2.1426. Epub 2022 Nov 9. PMID 36352489
- [Background] Driscoll A, Gao L, Watts JJ. Clinical effectiveness and cost-effectiveness of ambulatory heart failure nurse-led services: an integrated review. BMC Cardiovasc Disord. 2022 Feb 22;22(1):64. doi: 10.1186/s12872-022-02509-9. PMID 35193503
- [Background] De Maria M, Ausili D, Lorini S, Vellone E, Riegel B, Matarese M. Patient Self-Care and Caregiver Contribution to Patient Self-Care of Chronic Conditions: What Is Dyadic and What It Is Not. Value Health. 2022 Jul;25(7):1165-1173. doi: 10.1016/j.jval.2022.01.007. Epub 2022 Mar 23. PMID 35337754
- [Background] Chen J, Aronowitz P. Congestive Heart Failure. Med Clin North Am. 2022 May;106(3):447-458. doi: 10.1016/j.mcna.2021.12.002. Epub 2022 Apr 4. PMID 35491065
- [Background] Bas-Sarmiento P, Fernandez-Gutierrez M, Poza-Mendez M, Marin-Paz AJ, Paloma-Castro O, Romero-Sanchez JM; ASyAG_PPIC Team. Development and Effectiveness of a Mobile Health Intervention in Improving Health Literacy and Self-management of Patients With Multimorbidity and Heart Failure: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Apr 29;11(4):e35945. doi: 10.2196/35945. PMID 35486437
- [Background] Bas-Sarmiento P, Fernandez-Gutierrez M, Poza-Mendez M, Carrasco-Bernal MA, Cuenca-Garcia M, Diaz-Rodriguez M, Gomez-Jimenez MP, Paloma-Castro O, Torres-Castano A, Marin-Paz AJ. Needs of patients with multi-morbidity and heart failure for the development of a mHealth to improve their self-management: A qualitative analysis. Digit Health. 2023 Jun 8;9:20552076231180466. doi: 10.1177/20552076231180466. eCollection 2023 Jan-Dec. PMID 37325072
- [Background] Al-Hassan NM, Aldohaim SA, Benhjji MA, Al-Harbi OK, Alsaadi NA, Almogbel O, Elnour E, Hersi A. Prevalence and risk of hospitalization for depression in patients with heart failure. Curr Probl Cardiol. 2024 Nov;49(11):102793. doi: 10.1016/j.cpcardiol.2024.102793. Epub 2024 Aug 8. PMID 39122100
- [Background] Alconero-Camarero AR, -Romero AG, Sarabia-Cobo CM, Arce AM. "Clinical simulation as a learning tool in undergraduate nursing: Validation of a questionnaire". Nurse Educ Today. 2016 Apr;39:128-34. doi: 10.1016/j.nedt.2016.01.027. Epub 2016 Feb 4. PMID 27006044

DOCUMENTS (2):
  • Statistical Analysis Plan (2025-06-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT06855719/SAP_002.pdf
  • Informed Consent Form (2025-02-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT06855719/ICF_001.pdf